CLINICAL TRIAL: NCT06470893
Title: Online Exposure Therapy for Obsessive-Compulsive Disorder (OCD) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Kiara Timpano, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20240483
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OCD-NET Group (Experimental): Participants will receive the OCD-NET intervention for up to 12 months.
  Interventions: Behavioral: OCD-NET

INTERVENTIONS:
Behavioral: OCD-NET — OCD-NET is bibliotherapy with coaching and its content is reflective of standard care for OCD. OCD-NET is a self-paced intervention that participants complete entirely online with the support of an assigned individual therapist. Most participants complete this treatment in up to twelve weeks. On average, participants are expected to spend between one to five hours per week during the first half of treatment. In the second half of treatment when participants begin regular exposure and response prevention (ERP) exercises, participants are expected to spend about one hour per day.

SUMMARY:
The overarching goal of this protocol is to investigate mechanisms that influence symptom outcomes of exposure and response prevention (ERP) therapy for OCD. Mechanisms may include affective processes, learning factors, cognitive factors, or other constructs that could influence treatment outcomes. The study team will conduct this research within the context of an effective online treatment for OCD called OCD-NET. OCD-NET is bibliotherapy with coaching and its content is reflective of standard care for OCD.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Located within the United States
* 18-90 years old
* Able to provide consent
* Current diagnosis of OCD as assessed by clinical interview

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Participants currently located outside of the United States
* Prisoners
* Participants with hoarding as the primary OCD symptom
* Severe mental illness (e.g. schizophrenia, substance abuse); organic brain syndrome; or serious, current suicidal/homicidal ideation (based on phone screening or initial assessment)
* Concurrent enrollment in another psychotherapy treatment
* Participants taking psychotropic medication may be excluded if:

  * They have started a brand new psychotropic medication within the last 12 weeks
  * They have changed the dose of their psychotropic medication within the last 4 weeks
  * They anticipate that they cannot maintain the current dose of their psychotropic medication for the duration of the study
* Participants may be excluded if they have any cognitive or physical impairments that would interfere with their participation (e.g., significant head injury, cognitive disability, dementia).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Change in OCD Symptoms Measured by Yale-Brown Obsessive Compulsive Scale-Second Edition (YBOCS-II) | Baseline, up to 12 months (end of treatment)
  YBOCS-II scores range from 0-50, and higher scores indicate more severe illness

CONTACTS AND LOCATIONS:
Overall Officials: Kiara Timpano, PhD, Study Chair — University of Miami; Amelia Dev, MS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No